CLINICAL TRIAL: NCT03403933
Title: Study of the Effect of Calcifediol Supplementation on Left Ventricular Function in Cardiopathic Patients Undergoing Major Orthopedic Surgery
Brief Title: Vitamin D Supplementation on in Major Orthopedic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vitamina D (PI: M Turiel); L4073 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2017-12-19; First posted 2018-01-19 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Hypovitaminosis D; Cardiovascular Diseases
MeSH Terms: conditions — Vitamin D Deficiency; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cardiopathic patients in hypovitaminosis (Experimental): Didrogyl 10 ml: 10 drops a day to obtain levels of vitamin D > 30 ng /ml. Once these values are obtained lower the dose to 4-5 drops a day, with the aim, however, of keeping the plasma values between 30 and 60 ng/ml during 6 months of the study
  Interventions: Drug: Didrogyl

INTERVENTIONS:
Drug: Didrogyl — Calcifediol will be administered at a dose of 10 drops per day (as indicated for use) for 6 months or until vitamin D levels> 30 ng / ml are obtained.
  Once these values have been obtained, the dosage can be reduced to a dosage of 4/5 drops of calcifediol (1 drop contains 5mcg of calcifediol) with the aim to maintain the plasma values of 25 (OH) D in a optimal range between 30-60 ng / ml during the 6 month of the duration of the study.

SUMMARY:
Prospective, monocentric study in open, aimed at evaluating the effects of supplementation with calcifediol on left ventricular function parameters in cardiopathic subjects undergoing major orthopedic surgery.

DETAILED DESCRIPTION:
Population of the study: 47 cardiopathic patients with hypovitaminosis D supplemented with calcifediol to reach vitamin D levels> 30 ng / ml within 6 months. The purpose of this study is to evaluate the improvement of the ejection fraction or GLS (global longitudinal strain) calculated by speckle tracking at 6 months in cardiopathic patients with vitamin D deficiency during functional recovery after major orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: > or equal to 55 years, < or equal to 85 years
* cardiopathic patients (including hypertension) who must undergo major orthopedic surgery at our site
* patients with diagnosis: hypovitaminosis d

Exclusion Criteria:

* presence of neoplasm
* endocrinological pathologies excluding diabetes mellitus
* advanced chronic renal failure (GFR < 35 ml/min)
* pregnant women
* impossibility to participate to the rehabilitation protocol or to perform the established controls

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-09-23 (Actual); Study Completion 2018-07-16 (Actual)

PRIMARY OUTCOMES:
Evaluation of improvement of ejection fraction (FE) | 6 months
  Evaluation of improvement of ejection fraction (FE) or longitudinal strain calculated by speckle tracking at 6 months in cardiopathic patients with vitamin D deficiency who underwent supplementation with calcifediol, during functional recovery after major orthopedic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Turiel, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy